CLINICAL TRIAL: NCT00868140
Title: Determination if Indirectly Reducing Circulating Insulin by Improving Insulin Sensitivity With Pioglitazone Reduces Renal Clearance of D-chiro-inositol (DCI) Increases the Circulating Concentration of DCI and Enhances Insulin-stimulated Release of the D-chiro-inositol-containing Inositolphosphoglycan (DCI-IPG) Mediator in Obese Women With PCOS
Brief Title: Effects of Pioglitazone on Insulin and Glucose Metabolism in Women With Polycystic Ovary Syndrome (PCOS)
Acronym: PCOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: VCUIRB4480; GCRC0824 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1/Pioglitazone (Experimental): Pioglitazone in pill form at 45mg twice per day for 6 months
  Interventions: Drug: pioglitazone
- 2/Placebo (Placebo Comparator): Placebo control to arm 1 in pill form identical to treatment form also twice per day for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: pioglitazone — pioglitazone 45 mg
  Arms: 1/Pioglitazone
Drug: Placebo — placebo daily
  Arms: 2/Placebo

SUMMARY:
Our hypothesis is that hyperinsulinemia increases the renal clearance of D-chiro-inositol (DCI) in women with polycystic ovary syndrome (PCOS) and that this leads to a reduction in circulating insulin-stimulated D-chiro-inositol-containing inositol phosphoglycan (DCI-IPG) release. To assess the effects of a chronic reduction in circulating insulin on DCI metabolism, we propose to reduce circulating insulin in obese women with PCOS by improving insulin sensitivity with the drug pioglitazone. Pioglitazone is a thiazolidinedione that improves peripheral insulin sensitivity, presumably by activation of the peroxisome proliferator-activated receptor gamma (PPARγ) receptor. Administration of pioglitazone to women with PCOS has been shown to improve insulin sensitivity, reduce insulin secretion, and decrease both fasting and post-prandial serum insulin concentrations.

DETAILED DESCRIPTION:
This protocol focuses on the hypothesis that a deficiency in a putative inositolphosphoglycan (IPG) mediator of insulin action, namely a D-chiro-inositol-containing IPG (DCI-IPG), contributes to the insulin resistance of some women with PCOS. Our interest in this area stems directly from our previous studies, which demonstrated that administration of the precursor, D-chiro-inositol (DCI), to both obese and lean women with PCOS improved glucose intolerance while reducing circulating insulin, and simultaneously improved ovulatory function and decreased serum androgens. These findings were recently confirmed in a large-scale study by an independent group. The findings of these three studies suggested that administration of DCI improved insulin sensitivity in PCOS, which then resulted in an improved hormonal and metabolic milieu.

ELIGIBILITY:
Inclusion Criteria:

1. Obese (Body Mass Index or BMI greater than or equal to 30 kg/m2) women with PCOS between 18-40 years of age:

   * oligomenorrhea (less than 8 menstrual periods annually)
   * biochemical hyperandrogenemia (elevated total or free testosterone)
   * normal thyroid function tests and serum prolactin; AND
   * exclusion of 21a-hydroxylase deficiency by a fasting 17a-hydroxyprogesterone less than 200 ng/dl.51,
2. acceptable health on the basis of interview, medical history, physical examination, and laboratory tests (Complete Blood Chemistry or CBC, Comprehensive Metabolic Panel denoted SMA20, urinalysis, negative pregnancy test).
3. Signed, witnessed informed consent.
4. Ability to comply with study requirements.

Exclusion Criteria:

1. Diabetes mellitus by fasting glucose or oral glucose tolerance test (OGTT), or clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, neoplastic and malignant disease (other than non-melanoma skin cancer).
2. Current use of oral contraceptives.
3. Documented or suspected recent (within one year) history of drug abuse or alcoholism.
4. Ingestion of any investigational drug within two months prior to study onset.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Nestler, M.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- Virginia Commonwealth University General Clinical Research Center, Richmond, Virginia, United States
- Hospital de Clinical Caracas, Caracas, Venezuela

IPD SHARING:
Plan to Share IPD: No
individual data kept confidential, secured and not shared beyond authorized study staff

REFERENCES:
- [Result] Gupta A, Jakubowicz D, Nestler JE. Pioglitazone Therapy Increases Insulin-Stimulated Release of d-Chiro-Inositol-Containing Inositolphosphoglycan Mediator in Women with Polycystic Ovary Syndrome. Metab Syndr Relat Disord. 2016 Oct;14(8):391-396. doi: 10.1089/met.2016.0009. Epub 2016 Mar 30. PMID 27028341

RESULTS

PARTICIPANT FLOW:
Groups:
- 1/Pioglitazaone Treated: Pioglitazone treated subjects
  pioglitazone: pioglitazone 45 mg
- 2/Placebo: Placebo control to arm 1
  Placebo: placebo daily
Period: Overall Study
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Started | 26 | 25
Completed | 26 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 32 obese (body mass index, BMI, greater than or equal to 30 kg/m2 PCOS women, between 18-40 years old, were studied during the equivalent of the follicular phase of the menstrual cycle, as documented by a serum progesterone of less than or equal to 2 ng/ml.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Females | 16 | 16 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 19
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Venezuela | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: AUC DCI-IPG (%/Min)
Description: Change in the Area Under the Curve DCI-IPG measurements in blood samples taken at 15 minute intervals during the 2 hour OGTT before treatment with pioglitazone or placebo. Values reported as a percentage of bioactivity measured at time 0. Negative values indicate a decrease relative to the time 0 measurement.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: % bioactivity at time 0 of OGTT
Groups:
- 1/Pioglitazaone Treated: Pioglitazone
  pioglitazone: pioglitazone 45 mg
- 2/Placebo: control to arm 1
  Placebo: placebo daily
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
% bioactivity at time 0 of OGTT | 13162.06 (1240.6) | 14054.17 (1373.1)

2. Secondary Outcome: Matsuda Index
Description: Whole body insulin sensitivity as determined by the Matsuda Index as calculated using the following formula:
  10,000 divided by the square root of (FPI* FPG) * (xGPC* xIPC) Where FPI is fasting plasma insulin expressed as uU/ml, FPG is fasting plasma glucose expressed as mg/dL, xGPC is mean plasma glucose concentration after the load and xIPC is the mean insulin concentration after the load.
  Values calculated on samples taken at 0, 30, 60, 90 and 120 minutes of a 2 hour OGTT. Values typically range from 0 to 12 units with higher scores indicating better insulin sensitivity. A value of 2.5 or less is indicative of insulin resistance.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 3.36 (0.18) | 3.05 (0.15)

3. Primary Outcome: AUC DCI-IPG (%/Min)
Description: Change in the Area Under the Curve DCI-IPG measurements in blood samples taken at 15 minute intervals during the 2 hour OGTT following 6 months of treatment with pioglitazone or placebo. Values reported as a percentage of bioactivity measured at time 0. Negative values indicate a decrease relative to the time 0 measurement.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: % bioactivity at time 0 of OGTT
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
% bioactivity at time 0 of OGTT | -412.22 (1295.7) | -699.45 (1890.71)

4. Primary Outcome: Fasting Serum Insulin
Description: Fasting serum insulin (uIU.min/ml) measured at 0, 60 and 120 minutes of a 2 hour OGTT before treatment with either pioglitazone or placebo
Time Frame: baseline
Measure: Mean (Standard Error); unit: uIU.min/ml
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
uIU.min/ml | 15.04 (1.23) | 15.91 (1.32)

5. Primary Outcome: Fasting Serum Insulin (uIU/ml)
Description: Fasting serum insulin (uIU.min/ml) measured at 0, 60 and 120 minutes of a 2 hour OGTT following 6 months treatment with either pioglitazone or placebo
Time Frame: 6 months
Measure: Mean (Standard Error); unit: uIU.min/ml
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
uIU.min/ml | -8.69 (1.23) | -0.24 (1.50)

6. Secondary Outcome: Matsuda Index
Description: Whole body insulin sensitivity as determined by the Matsuda Index
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 1/Pioglitazaone Treated | 2/Placebo
Number analyzed (Participants) | 16 | 16
units on a scale | 4.29 (0.36) | 0.29 (0.17)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 1/Pioglitazone | 2/Placebo
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 3/26 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Pioglitazone (N=26) | 2/Placebo (N=25)
Edema (General disorders) | 3 (3) | 0 (0) — weight gain due to edema

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No